CLINICAL TRIAL: NCT05815667
Title: Effects of the Swedish Internet-based Individualised Active Communication Education (I-ACE) in First Time Hearing Aid Users: a Randomised Controlled Trial.
Brief Title: Effects of the Swedish Internet-based Individualised Active Communication Education (I-ACE) in FTU
Acronym: I-ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horselvarden Region Ostergotland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAK RCT
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): I-ACE. All participants are offered the I-ACE programme for the duration of 5 weeks.
  Interventions: Behavioral: Individualised Active Communication Education (I-ACE)
- Control group (No Intervention): Waiting list.

INTERVENTIONS:
Behavioral: Individualised Active Communication Education (I-ACE) — The swedish I-ACE consists of five modules with different themes, all with sections of information alternated with reflective tasks. The participants are assigned one module each week and provided with weekly feedback from a health care professional on their work, before being assigned the next module.
  Arms: Intervention group

SUMMARY:
Hearing impairment affects the ability to communicate, which can adversely affect both mental and physical health. The most common used rehabilitation method in hearing impairment is hearing aid fitting. Even with optimally fitted hearing aids, many struggle to hear in situations with difficult listening conditions. Active Communication Education (ACE) is an interactive group rehabilitation programme aiming to help those with hearing loss communicate more effectively using communication strategies to cope better in everyday life. An Individualised Active Communication Education (I-ACE) distributed digitally could enable those unable to get to the hearing care facility, or don't want to join the group sessions to benefit from the programme.

This project aims to investigate the effects of the swedish digital version of the I-ACE in first time hearing aid users.

ELIGIBILITY:
Inclusion Criteria:

* Adults >20 years old who have been fitted with hearing aids for the first time (first time users) 6 - 12 months prior.
* Computer experience and access to computer, tablet and/or smartphone with internet access.
* Access to BankID or equivalent.

Exclusion Criteria:

* Those who have participated in Active Communication Education prior.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Communication and Acceptance Scale (CAS) | Baseline, directly post intervention and 6 months post intervention.
  Assessing changes in use of communication strategies and the emotional consequences, knowledge and acceptance of hearing loss.
  Minimum 18 points to maximum 90. Higher score indicates a lower impact of the hearing loss.

SECONDARY OUTCOMES:
Communication Strategies Scale (CSS) | Baseline, directly post intervention and 6 months post intervention.
  Assessing changes in use of verbal, non-verbal and maladaptive communication strategies.
  Minimum 25 points to maximum 100. Higher score indicates a greater use of communication strategies.
The Hearing Handicap Inventory for the Elderly (HHIE) | Baseline, directly post intervention and 6 months post intervention.
  Assessing changes in emotional and social effects of hearing loss. Minimum 0 points to maximum 100 points. Higher score indicates greater emotional and social effects of hearing loss.
The International Outcome Inventory for Hearing Aids (IOI-HA) | Baseline, directly post intervention and 6 months post intervention.
  Assessing changes in perceived effectiveness and satisfaction with hearing aids.
  Minimum 7 points to maximum 35 points. Higher score indicates higher perceived effect.
The International Outcome Inventory for Alternative Interventions (IOI-AI) | Directly post intervention and 6 months post intervention.
  Assessing changes in perceived effectiveness with an alternative intervention, in this case the I-ACE.
  Minimum 7 points to maximum 35 points. Higher score indicates higher perceived effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Hörselvården Region Östergötland, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No